CLINICAL TRIAL: NCT05274373
Title: Clinical, Virological, Serological and Immunological Characteristics During and Following COVID-19 Hospitalization: a Prospective Cohort Study
Brief Title: Clinical, Virological, Serological and Immunological Characteristics During and Following COVID-19 Hospitalization
Acronym: COVISERA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Statens Serum Institut (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: Covisera
Record Dates: First submitted 2022-03-08; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pneumonia; COVID-19
Keywords: Neutralizing Antibodies; Viral Load; Antibody Decay; Viral Culturing; Infectiousness
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — 1. Oropharyngeal swabs
  2. Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the association between the severity of COVID-19 and SARS-CoV-2 NAb titers levels for up to six months following primary infection using a live virus NAb assay. Description of SARS-CoV-2 viral shedding and infectiousness during the first 30 days after infection in a group of unvaccinated hospitalized patients.

DETAILED DESCRIPTION:
The studys primary aim is to assess clinical factors, such as disease severity, associated with neutralizing antibody (NAb) production. Furthermore, the study aims to assess the length of SARS-CoV-2 infectiousness and clinical factors associated with viral load.

Patients 18 years or older hospitalized at Copenhagen University Hospital at North Zealand, Copenhagen, Denmark, May 24th,2020 - May 5th, 2021, were routinely screened for COVID-19 by diagnostic oropharyngeal or tracheal RT-PCR samples taken during admission. Patients with a positive SARS-CoV-2 PCR within 48 hours from hospital admission were offered inclusion, if COVID-19 pneumonia was confirmed.

The following were retrieved from patients' electronic records: comorbidities (Charlson Comorbidity Index),vital signs (Early Warning Score), immunocompromised status, time from symptom onset to admission, oxygen treatment, pharmacological treatment, admission length, death and bacterial co-infection.

Paired oropharyngeal swabs and serum samples were collected at inclusion (day 0), days 3, 7, 10, 14, 17, 24, and 30. Serum samples were, if possible, also collected after three and six months. Follow-up time was six months.

RT-qPCR analysis targeted the SARS-CoV-2 RNA-dependent-RNA-polymerase (RdRp)-helicase gene region and two samples with known viral load were included in each PCR-run for quantification of patient samples. Virus was cultured in African green monkey cells (VERO-E6) with incubation for 3 - 4 days and daily microscopic inspection for cytopathogenic effect (CPE). A total of three passages were made before the the virus was interpreted as non-replicant. Cells with CPE were confirmed by RT-qPCR.

The presence of specific antibodies (Ab) against SARS-CoV-2 in serum was assessed using Wantai total-Ab ELISA according to the manufacturer's instructions (Wantai, Beijing, China).

For the in-house live virus NAb analysis, a 50% cut-off value was calculated from quadruplicate virus and cell control wells included on each plate using the following equation: (average optical density (OD) of virus control wells + average OD of cell control wells)/2. The 50% neutralization titer was calculated as the interpolation of the cutoff value with a four-parameter logistic regression curve fitted for each serum serial dilution. To minimize inter-assay variation, the titers were normalized according to a positive control included on each assay plate.

A linear mxied-effects model was used to assess the association between repeated NAb measurements and clinical variables such as age, gender and disease severity. A linear mixed-effects model was also used to assess the association between repeated viral load measurements and clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* positive SARS-CoV-2 specimen from upper or lower respiratory tracts (virological criteria)
* consolidations on the chest X-ray described by a radiologist, treating physician or a physician from the study group (radiological criteria)
* the presence of one or more of the following: fever (temperature ≥38.0°C), new-onset cough, pleuritic chest pain, dyspnea or altered breath sounds on auscultation (clinical criteria)

Exclusion Criteria:

* cognitive impairment prohibiting giving informed consent to participation
* by December 14th, 2020, and onwards patients if the time since symptom onset was > seven days at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult unvaccinated hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-05-24 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Neutralizing Antibody Titer - Day 0 | Day 0
  Baseline Log10 Spike protein neutralizing antibody titer
Change from baseline in Neutralizing Antibody Titer - Day 30 | Day 30
  Log10 Spike protein neutralizing antibody titer
Change from baseline in Neutralizing Antibody Titer - Day 90 | Day 90
  Log10 Spike protein neutralizing antibody titer
Change from baseline in Neutralizing Antibody Titer- Day 180 | Day 180
  Log10 Spike protein neutralizing antibody titer
Viral culturing - Day 0 | Day 0
  Number of successful viral culturing attempts (SARS-CoV-2)
Viral culturing - Day 3 | Day 3
  Number of successful viral culturing attempts (SARS-CoV-2)
Viral culturing - Day 7 | Day 7
  Number of successful viral culturing attempts (SARS-CoV-2)
Viral culturing - Day 10 | Day 10
  Number of successful viral culturing attempts (SARS-CoV-2)
Viral culturing - Day 14 | Day 14
  Number of successful viral culturing attempts (SARS-CoV-2)
Viral culturing - Day 17 | Day 17
  Number of successful viral culturing attempts (SARS-CoV-2)
Viral culturing - Day 24 | Day 24
  Number of successful viral culturing attempts (SARS-CoV-2)
Viral culturing - Day 30 | Day 30
  Number of successful viral culturing attempts (SARS-CoV-2)

SECONDARY OUTCOMES:
Baseline Viral Load - Day 0 | Day 0
  Log10 copies/ml
Change from Baseline Viral Load - Day 3 | Day 3
  Log10 copies/ml
Change from Baseline Viral Load - Day 7 | Day 7
  Log10 copies/ml
Change from Baseline Viral Load - Day 10 | Day 10
  Log10 copies/ml
Change from Baseline Viral Load - Day 14 | Day 14
  Log10 copies/ml
Change from Baseline Viral Load - Day 17 | Day 17
  Log10 copies/ml
Change from Baseline Viral Load - Day 24 | Day 24
  Log10 copies/ml
Change from Baseline Viral Load - Day 30 | Day 30
  Log10 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: Zitta Barrella Harboe, MD, PhD, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Copenhagen University Hospital at North Zealand, Copenhagen, Denmark

REFERENCES:
- [Derived] Sejdic A, Frische A, Jorgensen CS, Rasmussen LD, Trebbien R, Dungu A, Holler JG, Ostrowski SR, Eriksson R, Soborg C, Nielsen TL, Fischer TK, Lindegaard B, Franck KT, Harboe ZB. High titers of neutralizing SARS-CoV-2 antibodies six months after symptom onset are associated with increased severity in COVID-19 hospitalized patients. Virol J. 2023 Jan 25;20(1):14. doi: 10.1186/s12985-023-01974-8. PMID 36698135